CLINICAL TRIAL: NCT07111325
Title: A Clinical Trial Study Evaluating the Safety and Preliminary Efficacy of Human Induced Pluripotent Stem Cell-derived Extracellular Vesicles (iEVs) Injection for the Treatment of Lateral Epicondylitis of the Humerus
Brief Title: Safety and Preliminary Efficacy of iEVs Injection in Treating Lateral Epicondylitis of Humerus
Acronym: iEVs
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Jian Ding, Doctor, Shanghai 6th People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-052
Record Dates: First submitted 2025-07-31; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Lateral Epicondylitis
Keywords: lateral epicondylitis; tennis elbow; induced pluripotent stem cell; extracellularvesicles
MeSH Terms: conditions — Tennis Elbow | interventions — Immobilization

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- iEV-high (Experimental): 1X10^10/ml
  Interventions: Biological: iEV; Other: immobilization
- iEV-Low (Experimental): 1X10^9/ml
  Interventions: Biological: iEV; Other: immobilization
- PRP (Active Comparator): PRP
  Interventions: Biological: PRP; Other: immobilization
- Control (Other)
  Interventions: Other: immobilization

INTERVENTIONS:
Biological: iEV — induced pluripotent stem cell-derived extracellular vesicles
  Arms: iEV-Low; iEV-high
Biological: PRP — PRP injection
  Arms: PRP
Other: immobilization — immobilization

SUMMARY:
Evaluate the safety and preliminary efficacy of human induced pluripotent stem cell-derived extracellular vesicle (iEV) injection in the treatment of lateral epicondylitis of the humerus.

DETAILED DESCRIPTION:
Lateral epicondylitis refers to pain at the lateral epicondyle of the humerus caused by chronic traumatic tendinopathic changes in the origin and insertion of the common extensor tendon on the lateral side of the elbow joint, which result from long-term and repeated loading.

This randomized controlled study aims to observe whether extracellular vesicles derived from human induced pluripotent stem cells (iEVs) can promote the improvement of inflammatory status in injured extensor tendons and alleviate clinical symptoms. The study design will evaluate the efficacy by assessing changes in patients' pain, grip strength, and elbow joint function after treatment with the injection, and compare the efficacy with that of the control groups.

This is an interventional, single-center clinical study. The study plans to adopt a block randomization method without stratification. A randomization list will be generated separately for each research center by a computer, and participants will be randomly assigned to the experimental group, positive control group, and negative control group. There will be 6-12 cases in the experimental group, and 3-6 cases in each of the two control groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with lateral epicondylitis by clinical symptom examination and MRI or ultrasound, without obvious tendon tear;
* Unilateral lateral elbow pain lasting for more than 12 weeks;
* Pain is provoked by at least 2 of the following methods, with a pain VAS score exceeding 3: maximum grip strength, palpation of the lateral epicondyle of the elbow and surrounding area, resisted dorsiflexion of the wrist or middle finger, or stretching of the forearm extensor muscles under a pain-free grip state;
* Having received physical therapy or non-steroidal anti-inflammatory drug treatment with poor efficacy;
* Individuals with independent behavioral capacity, who have signed the informed consent form themselves.

Exclusion Criteria:

* Complaints of ipsilateral muscle pain caused by other reasons in the past 6 months;
* Presence of ipsilateral neurogenic, inflammatory, or systemic joint diseases;
* A history of previous lateral epicondylitis (LET) surgery in the past 6 months;
* Subjects deemed unsuitable for participating in the trial due to other conditions, as judged by the researcher;
* MRI showing that the injury has involved the lateral collateral ligament, with concurrent cartilage damage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess changes in pain levels using a Visual Analogue Scale (VAS) | From enrollment to the end of treatment at 12 weeks
  Assess changes in pain levels using the Visual Analogue Scale (VAS). The scale ranges from 0 (no pain) to 10 (the most severe pain), where a higher score indicates more severe pain (worse outcome) and a lower score indicates less severe pain (better outcome).
Evaluate changes in functional outcomes through patient-rated tennis elbow assessments (PRTEE) | From enrollment to the end of treatment at 12 weeks
  To assess changes in functional outcomes, the Patient-Rated Tennis Elbow Evaluation (PRTEE) is utilized. This scale encompasses 15 items, divided into two dimensions: the pain dimension (5 items) and the function dimension (10 items). It uses a 0-10 scoring system, where a higher total score indicates more severe functional impairment (worse outcome), and a lower total score indicates less severe functional impairment (better outcome).
Assess changes in functional outcomes using the Mayo Elbow Performance Score (MEPS) | From enrollment to the end of treatment at 12 weeks
  To assess changes in elbow function, the Mayo Elbow Performance Score (MEPS) is employed. This scale ranges from 0 to 100, where a higher score indicates better elbow function (better outcome) and a lower score indicates worse elbow function (worse outcome).
Incidence of adverse events | From enrollment to the end of treatment at 12 weeks

SECONDARY OUTCOMES:
Changes in the results of the SF-36 Quality of Life Questionnaire | From enrollment to the end of treatment at 12 weeks
Changes in functional outcomes assessed by the Subjective Elbow Value (SEV) | From enrollment to the end of treatment at 12 weeks
MRI imaging assessment at 3 months after injection | From enrollment to the end of treatment at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth hospital, Shanghai, Shanghai Municipality, China